CLINICAL TRIAL: NCT00431626
Title: A Randomized, Placebo-Controlled, Double-Masked Clinical Trial Comparing Laser TURP With and Without Neo-Adjuvant Dutasteride
Brief Title: A Clinical Trial Comparing Laser TURP With and Without Dutasteride.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Northwestern University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Kevin McVary, Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0348-040
Record Dates: First submitted 2007-02-02; First posted 2007-02-06 (Estimated); Results first posted 2015-01-01 (Estimated); Last update posted 2015-10-28 (Estimated); Status verified 2015-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Benign; Prostatic; Hyperplasia; Lower; Urinary; Track; Symptoms; Laser; Transurethral; Prostate
MeSH Terms: conditions — Prostatic Hyperplasia; Hyperplasia | interventions — Dutasteride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laser TURP with dutasteride (Experimental): Prior to and after standard treatment with laser TURP, dutasteride is applied to each patient
  Interventions: Drug: Dutasteride (Avodart)
- Laser TURP with placebo (Placebo Comparator): Prior to and after standard treatment with laser TURP, placebo is applied to each patient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dutasteride (Avodart)
  Arms: Laser TURP with dutasteride
Drug: Placebo — Placebo before and after treatment of TURP
  Arms: Laser TURP with placebo

SUMMARY:
The purpose of this research study is to determine if the study drug Dutasteride taken before and after Laser TURP(Transurethral Resection of the Prostate), can provide effective and safe, long term improvement of lower urinary tract symptoms.

DETAILED DESCRIPTION:
Benign Prostatic Hyperplasia (BPH) is the most common neoplastic condition afflicting middle-aged and elderly men. BPH is a non-cancerous condition in which the prostate becomes enlarged which can cause lower urinary tract symptoms (LUTS). These symptoms include: frequency, urgency, weak urinary stream, difficulty starting or stopping to urinate and feeling the need to urinate even after just finishing urinating.

One of the minimally invasive treatments for BPH is a Laser TURP. The men going into this study would be planning on having a Holmium Laser TURP at Northwestern Memorial Hospital in Chicago, Illinois.

Another treatment for BPH is the use of a class of drugs called 5-Alpha Reductase Inhibitors (5ARI). Dutasteride is a 5ARI that has been approved by the U.S. Food and drug Administration (FDA) for the treatment of BPH.

Each participant in this study will be randomized into ONE of the treatment groups below:

1. Laser TURP combined with Dutasteride
2. Laser TURP combined with placebo.

This study is double-masked which means neither the participant, nor the study staff will know who is receiving active study drug or placebo. There will be a 50% chance of receiving the study drug, Dutasteride, and a 50% chance of receiving a placebo.

Dutasteride or it's placebo comes as a 0.5mg capsule to be taken by mouth once a day at bedtime.

There will be a screening period that may last up to 8 weeks. It will include:

* There will be 2 or 3 screening visits to the clinic with each visit lasting approximately 2.5 to 3 hours.
* Each participant will be asked to complete various forms and questionnaires regarding their lower urinary tract symptoms and how they effect them and their sexual function.
* No study drug will be taken during this time.
* The Laser TURP at Northwestern Memorial Hospital will be scheduled.

If each requirement has been met and it is determined that the participant is eligible to participate in this trial the participant will come to the clinic for a randomization visit.

At this visit the participant will be randomized into one of the two treatment groups noted above. Randomization is like a flip of a coin and neither the participant, nor the study staff chooses which treatment will be given.

Each participant will start taking the study drug everyday for six weeks before undergoing the Laser TURP and will continue taking the study drug every day for one year after the Laser TURP.

If the Laser TURP requires having a catheter in place, the participant will be seen by the urology clinic staff for follow up visits for this catheter. This follow up schedule may require weekly visits.

There will be follow up visits with the research staff. The participant will be asked to come to the research clinic every three months for one year. Each follow up visit will last approximately 1.5 hours.

A final visit will take place at one year. This will be identical to the first screening visit. This visit will last approximately 2 hours.

If the participant decides to withdraw from this study early he will be asked to come into the office for an early withdrawal visit.

Please note: The above detailed information regarding this research study is not in it's entirety. All of the above and more will be discussed in complete detail upon meeting with a research staff member or by calling the contact person mentioned in this protocol registration below.

ELIGIBILITY:
Inclusion Criteria:

* The patient is a male at least 50 years of age.
* The patient's peak urinary flow rate is at least 4 ml/sec, but not greater than 15 ml/sec, and the voided volume is at least 125 ml.
* Prostate volume must be greater than 30 grams
* The AUA-SI is greater than or equal to 9.
* Patient must be scheduled for a Laser TURP or eligible to be scheduled for Laser TURP
* Patient must be able to complete the study requirements prior to the scheduled laser TURP.
* The patient has signed the informed consent prior to the performance of any study procedures.

Exclusion Criteria:

* The patient has had any prior surgical intervention for BPH.
* The patient is receiving any intervention for prostate disease (either medical or surgical) or is presently enrolled in any study protocol.
* The patient has had a previous hypersensitivity, idiosyncrasy, or clinically suspected drug reaction to dutasteride.
* The patient has taken an alpha-1 blocker within 1 month of randomization.
* The patient has taken finasteride or dutasteride within 3 months of randomization.
* The patient has taken phenylephrine, pseudoephedrine, imipramine, and an anticholinergic or cholinergic medication within 4 weeks of the screening visit.
* The patient has taken an estrogen, androgen, or any drug producing androgen suppression, or anabolic steroids.
* The patient has an inability to urinate.
* The patient has clinically significant renal or hepatic impairment (i.e., creatinine greater than 2.0 mg/dl or AST greater than 1.5 times the upper limit of normal).
* The patient has a PSA level greater than 10 ug/ml (Hybritech).
* The patient requires the daily use of a pad or device for incontinence.
* The patient has had an episode of unstable angina pectoris, a myocardial infarction, transient ischemic attack, or a cerebrovascular accident within the past six months.
* The patient has a penile prosthesis or artificial urinary sphincter.
* The patient has a history or current evidence of carcinoma of the prostate or bladder, pelvic radiation or surgery, urethral stricture, prior surgery for BPH, or bladder neck obstruction.
* The patient has an active urinary tract disease or has undergone cystoscopy or biopsy of the prostate within two weeks prior to the first screening visit.
* The patient has known primary neurologic conditions such as multiple sclerosis or Parkinson's disease or other neurological diseases known to affect bladder function.
* The patient has had documented bacterial prostatitis within the past year.
* The patient has had two documented urinary tract infections of any type in the past year. A urinary tract infection is defined as >100,000 colonies per ml urine from midstream clean catch or catheterized specimen.
* The patient has a severe bleeding disorder that makes laser TURP impossible.
* The patient must be able to stop any anticoagulant, NSAID or anti-platelet for 7 days prior to the laser TURP.
* The patient has had cancer that is not considered cured (except basal cell or squamous cell carcinoma of the skin). A patient is considered cured if there has been no evidence of cancer within five years of randomization.
* The patient has a diagnosis of a thought disorder (i.e., schizophrenia, bipolar disorder)
* The patient has any serious medical condition likely to impede successful completion of the study.
* The patient has a defibrillator that cannot be deactivated during laser TURP treatment.
* A bladder neck to verumontanum distance which is less than 30mm in length as measured by flexible cystoscopy and a total prostate volume <25 ml or >110 ml as measured by prostate volume ellipsoid formula during TRUS.

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2006-10; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin T. McVary, MD, Principal Investigator — Northwestern University

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 4 | 0
Completed | 4 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Laser TURP With Dutasteride: Prior to and after standard treatment with laser TURP, dutasteride is applied to each patient
  Dutasteride (Avodart)
- Total: Total of all reporting groups
Arm/Group | Laser TURP With Dutasteride | Laser TURP With Placebo | Total
Number analyzed (Participants) | 4 | 0 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 47 (12) |  | 47 (12)
Gender [Number; unit: participants]
  Female | 0 |  | 0
  Male | 4 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Measure Will be the 5 Point Change in AUA Symptom Index
Description: AUA symptoms index change is measured on a five level-scale: -2 (much worse), -1(worse) , 0 (no change), 1 (better), 2 (much better)
Time Frame: one year
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Laser TURP With Dutasteride | Laser TURP With Placebo
Number analyzed (Participants) | 4 | 0
units on a scale | 1 (0.8) |

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Laser TURP With Dutasteride | Laser TURP With Placebo
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/0
Other Adverse Events (participants affected / at risk) | 0/4 | 0/0

LIMITATIONS AND CAVEATS:
Difficulty in recruitment forced the closing of this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No